CLINICAL TRIAL: NCT05474001
Title: Intrathecal Fentanyl Versus Intravenous Granisetron for the Prevention of Perioperative Nausea and Vomiting During Cesarean Delivery Under Spinal Anesthesia
Brief Title: Comparison Between IT Fentanyl and IV Granisetron in Prevention of Vomiting in CS Under Spinal Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mohamed Youssef Mohamed (Other)
Responsible Party: Sponsor-Investigator, Mohamed Youssef Mohamed, Principal Investigator, Sohag University
Organization: Sohag University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 134896646
Record Dates: First submitted 2022-06-24; First posted 2022-07-26 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Nausea and Vomiting, Postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Fentanyl; Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fentanyl group (Active Comparator): Patients will receive 10 mg hyperbaric Bupivacaine ( 2ml ) and 20 μg (0.5 mL) fentanyl IT.
  1 mL IV normal saline immediately after the placement of the spinal.
  Interventions: Drug: Fentanyl
- Granisetron group (Active Comparator): Patients will receive 10 mg hyperbaric Bupivacaine ( 2ml ) and 0.5 mL normal saline IT.
  1 mg (1 mL) IV granisetron after spinal placement.
  Interventions: Drug: intravenous graniseton
- Control group (Placebo Comparator): 10 mg hyperbaric Bupivacaine ( 2ml ) IT and normal saline 0.5 ml
  1 ml normal saline IV after spinal placement.
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Fentanyl — 10mg bubivacain intrathecal ( 2ml ) with 20microgram intrathecal fentanyl
  Other Names: IT Fentanyl
  Arms: Fentanyl group
Drug: Bupivacain — 10mg bubivacain intrathecal (2ml) with 0.5 ml saline with no intrathecal fentanyl
  Other Names: IT mercaine
  Arms: Control group
Drug: intravenous graniseton — 10mg bubivacain intrathecal ( 2ml ) with 0.5 ml saline with no intrathecal fentanyl with 1mg iv granisetron
  Other Names: IV Grantryl
  Arms: Granisetron group

SUMMARY:
Intrathecal Fentanyl Versus Intravenous Granisetron for the Prevention of Perioperative Nausea and Vomiting During Cesarean Delivery under Spinal Anesthesia

DETAILED DESCRIPTION:
This prospective randomized control study will be held in Sohag University Hospital After approval of local ethics committee of sohag university hospital from June 2022 to December 2022, written informed consent will be taken from all patients , about advantages and possible complications of this study .

Inclusion criteria This study will include 90 Patients , physical status I or II according to ASA classification , age between ( 18 - 45 years ) undergoing cesarean delivery under spinal anesthesia.

Technique :

On arrival of patient to operative room :

1. 20G IV line ( cannula ) will be inserted .
2. Putting of patient on monitor and assessment of hemodynamics ( HR , RR , BP ) .
3. Pre anesthetic hydration by at least 1000 ml ringer lactate
4. Patient received Spinal anesthesia at level L3-L4 or L4-L5 lumbar segement .
5. during the procedure, If patient suffer from :

   * brady cardia with heart rate ( HR ) less than 55 we will give atropine sulphate 0.5 mg IV .
   * hypotension less than 25% of MBP of preoperative value we will give normal saline or ephedrine 5-10 mg .
6. Putting patient in the position for the operation .

Patients will be prospectively randomized divided into 3 groups :

The patients will be randomized using closed envelope method and the medications will be prepared by another anaesthologist not sharing in the study

Group ( F ) Fentanyl group : ( n = 30 ) Patients will receive 10 mg hyperbaric Bupivacaine ( 2ml ) and 20 μg (0.5 mL) fentanyl IT.

1 mL IV normal saline immediately after the placement of the spinal. Group ( G ) Granisetron group : ( n = 30 ) Patients will receive 10 mg hyperbaric Bupivacaine ( 2ml ) and 0.5 mL normal saline IT.

1 mg (1 mL) IV granisetron after spinal placement. Group ( C ) Control group : ( n = 30 ) 10 mg hyperbaric Bupivacaine ( 2ml ) IT and normal saline 0.5 ml

1 ml normal saline IV after spinal placement.

\Data will be collected from this study : ( 1 ) : Demographic data : Age , sex , weight , height and duration of operation .

( 2 ) : intraoperative:

A- hemodynamics (HR , BP , RR , oxygen saturation before anesthesia , after induction and then :

Every 5 minutes for 1st hour Every 15 minutes for next 2 hours Then every 3 hour for 12 h post operative . B - nausea and vomiting. C - patient discomfort during anesthesia. D - itching. ( 3 ) : post operative : A - nausea and vomiting : using nausea and vomiting score. B - pain assessment using VAS : every 30 mins for 2 h , every hour for 12 h If VAS 3-5 we will give paracetamol 1g IV , more than 5 we will give ketrolac 30 mg IV C _ total analgesic consumption D _ itching F _ retention of urine

ELIGIBILITY:
Inclusion Criteria:

* physical status I or II according to ASA classification with age between ( 18 - 45 years ) undergoing cesarean delivery under spinal anesthesia.

Exclusion Criteria:

* patient refusal .
* Any contraindication of neuraxial block.
* Patients with physical status other than 1 and 2 according to ASA classification
* Those with history of nausea and vomiting as Parturients with a history of motion sickness, hyperemesis gravidarum , also those who received anti emetic drugs in last 2 hours of operation .
* Allergy to any of the drug included in this study .
* complicated pregnancy as placenta previa, preeclampsia and eclampsia multible pregnancy
* fetal distress

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women undergoing cesarean section
Enrollment: 90 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
nausea and vomiting score in patient during caesarean delivery | six month
  : To compare intrathecal (IT) fentanyl with IV granisetron for preventing intraoperative nausea and vomiting during cesarean deliveries performed with spinal anesthesia.
  according to nausea and vomiting scale ( from 0 = no nausea , to 10= resistant nausea and vomiting )

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Intrathecal Fentanyl Is Superior to Intravenous Ondansetron for the Prevention of Perioperative Nausea During Cesarean Delivery with Spinal Anesthesia — https://journals.lww.com/anesthesia-analgesia/fulltext/2000/05000/intrathecal_fentanyl_is_superior_to_intravenous.30.aspx